CLINICAL TRIAL: NCT03990831
Title: Frontal Lobe Oxyhemoglobin Levels in Patients With Lower Extremity Burns Assessed Using a Functional Near-Infrared Spectroscopy Device During Usual Walking: A Pilot Study
Brief Title: Frontal Lobe Oxyhemoglobin Levels in Patients With Lower Extremity Burns Assessed Using a fNIRS
Acronym: fNIRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hangang Sacred Heart Hospital (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, So Young Joo, Department of Rehabilitation Medicine, Hangang Sacred Heart Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HangangSHH-1
Record Dates: First submitted 2019-02-21; First posted 2019-06-19 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Walking
Keywords: Burn; Near-infrared spectroscopy (NIRS)
MeSH Terms: conditions — Burns

STUDY DESIGN:
Intervention Model Description: patients with lower extremity burn : 15 patients patients with upper extremity burn : 10 patients healthy controls : 11
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- burn injury and normal patient (Other): HbO2 PFC perfusion using fNIRS
  Interventions: Diagnostic Test: Functional near-infrared spectroscopy (fNIRS)

INTERVENTIONS:
Diagnostic Test: Functional near-infrared spectroscopy (fNIRS) — Functional near-infrared spectroscopy (fNIRS) measurement

SUMMARY:
Investigators investigate the patterns of cortical activation using the NIRST in patients with peripheral neurological injury caused by lower extremity burns.

DETAILED DESCRIPTION:
Understanding the mechanisms associated with locomotor networks may be of benefit for rehabilitation of burn victims with neurological locomotor deficits. However, the effects of peripheral neurological injury on locomotor network remains unknown. A wearable functional near-infrared spectroscopy (fNIRS) device has been developed for studying cortical hemodynamics. Changes in cortical activity has not previously been documented in patients with burn injury.

Investigators assessed 15 patients with lower extremity burns and 11 healthy controls.

Investigators measured walking-related cortical activity using an fNIRS device at baseline and during usual walking.

Cortical activity was measured by evaluating relative changes in oxyhemoglobin level. The NIRST Analysis Tool v2.1 was utilized to analyze fNIRS data in a MATLAB environment.

ELIGIBILITY:
Inclusion Criteria:

* burn patients with lower extremity or upper extremity thermal injury
* patients who could walk unassisted for at least 5min.

Exclusion Criteria:

* patients with critical systemic conditions
* severe cognitive impairment
* had severe pain
* unable to walk.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2019-07-09 (Actual)

PRIMARY OUTCOMES:
oxygenated hemoglobin (HbO2) of the prefrontal regions, | 5 minutes
  identify the location of the normal cortical activation during usual walking

CONTACTS AND LOCATIONS:
Overall Officials: Cheong Hoon Seo, M.D., Principal Investigator — Hangang Sacred Heart Hospital
Locations (1):
- Hangang Sacred Heart Hospital, Seoul, Yeongdeungpo-Ku, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Yahya E, Johansen-Berg H, Kischka U, Zarei M, Cockburn J, Dawes H. Prefrontal Cortex Activation While Walking Under Dual-Task Conditions in Stroke: A Multimodal Imaging Study. Neurorehabil Neural Repair. 2016 Jul;30(6):591-9. doi: 10.1177/1545968315613864. Epub 2015 Oct 21. PMID 26493732
- [Background] Kim HY, Kim EJ, You JSH. Adaptive locomotor network activation during randomized walking speeds using functional near-infrared spectroscopy. Technol Health Care. 2017 Jul 20;25(S1):93-98. doi: 10.3233/THC-171310. PMID 28582896